CLINICAL TRIAL: NCT00000116
Title: Clinical Trial of Docosahexaenoic Acid (DHA) in Patients With Retinitis Pigmentosa Receiving Vitamin A Treatment
Brief Title: Randomized Trial of DHA for Retinitis Pigmentosa Patients Receiving Vitamin A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Carol Weigel DiFranco (NIH)
Responsible Party: Sponsor-Investigator, Carol Weigel DiFranco, coauthor/program manager, National Eye Institute (NEI)
Organization: National Eye Institute (NEI) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NEI-12
Record Dates: First submitted 1999-09-23; First posted 1999-09-24 (Estimated); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa | interventions — Vitamin A; Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In this trial neither the participants, nor the clinicians, nor the investigators were aware of treatment group assignment.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Docosahexaenoic acid + Vitamin A (Experimental): Participants randomized to this arm received 1200 mg/d docosahexaenoic acid and 15000 IU/d Vitamin A as retinyl palmitate
  Interventions: Dietary Supplement: Vitamin A; Dietary Supplement: Docosahexaenoic acid
- Control fatty acid + Vitamin A (Placebo Comparator): Patients randomized to this arm received 500 mg/d of fatty acid with no docosahexaenoic acid and 15000 IU/ Vitamin A as retinyl palmitate
  Interventions: Dietary Supplement: Vitamin A; Dietary Supplement: Control fatty acid

INTERVENTIONS:
Dietary Supplement: Vitamin A — 15000 IU/d as retinyl palmitate
Dietary Supplement: Docosahexaenoic acid — 1200 mg/d
  Arms: Docosahexaenoic acid + Vitamin A
Dietary Supplement: Control fatty acid
  Arms: Control fatty acid + Vitamin A

SUMMARY:
The purpose of this trial is to determine whether a nutritional supplement in addition to vitamin A will slow the course of retinitis pigmentosa.

DETAILED DESCRIPTION:
Retinitis pigmentosa (RP) is a group of inherited retinal degenerations with a worldwide prevalence of approximately 1 in 4,000. Patients typically report night blindness and difficulty with midperipheral visual field in adolescence. As the condition progresses, they lose far peripheral visual field. Most patients have reductions in central vision by age 50 to 80 years. Based on electroretinograms (ERGs), the course of the disease can be slowed on average among adults on 15,000 IU/day of vitamin A palmitate. While conducting the trial on the effects of vitamin A on RP, it became apparent that another substance in the diet could be affecting the course of the disease. This prompted the present randomized, controlled trial.

This study is a randomized, controlled, double-masked trial with a planned duration of 5 years. Patients with the common forms of RP are assigned to either a test or a control group. All receive 15,000 IU/day of vitamin A palmitate in addition to either 1200 mg/d of docosahexaenoic acid or control capsules. Participants will not know the contents of the supplement or the group to which they have been assigned until the end of the trial. The main outcome measurement is the total point score on the Humphrey Field Analyzer (HFA). In addition, computer-averaged 30-Hz cone ERG amplitudes and visual acuity are measured annually.

ELIGIBILITY:
Inclusion Criteria:

Ocular Criteria:

Retinitis Pigmentosa, typical (non-syndromic) forms Best corrected visual acuity Greater than or equal to (GE )20/100 HFA 30-2 total point score GE 250 dB (decibels) 30 (Hertz) Hz ERG cone amplitude GE 0.68 microvolts

Dietary Criteria:

Dark fish intake Less than or equal to (LE) five servings per week Dietary omega-3 fatty acid intake LE 0.41 g/d Preformed Vitamin A intake in diet and supplements LE 10,000 IU/d Supplement intake LE 5000 IU/d of Vitamin A and LE 30 IU/d Vitamin E Consumption LE 3 alcoholic beverages per day

Medical and other criteria:

Body Mass Index Less than (LT )40 and weight GE 5th percentile for age, sex, and height Serum retinol level LE 100 mg/dl and serum retinyl ester levels LE 380 nm/L Serum cholesterol level LT 300 mg/dL and serum triglyceride levels LT 400 mg/dL Agree not to know study capsule content

Exclusion criteria:

Ocular criteria:

No confounding ocular disease

Dietary criteria:

No intake of cod liver oil or omega-3 capsules

Medical and other criteria:

Not pregnant or planning to become pregnant No clinically significant abnormal result on Complete Blood Count or serum liver function profile No other disease which might affect absorption or metabolism of DHA or Vitamin A

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 221 (Actual)
Dates: Start 1996-05 (Actual); Primary Completion 2002-09 (Actual); Study Completion 2002-09 (Actual)

PRIMARY OUTCOMES:
Change in Humphrey Field Analyzer (HFA) total point score 30-2 program | Annual percent change per year at each of 4 years of followup
  Sum of points in Decibels of total points seen in 30-2 program. Higher scores = better vision/larger visual field

SECONDARY OUTCOMES:
Change in Humphrey Field Analyzer (HFA) total point score 30 -2 plus 30/60-2 programs combined | Annual percent change per year at each of four years of followup
  Sum of points in decibels of total points seen in 30-2 and 30/60-2 programs combined- Higher scores = better vision/ larger visual field
Change in 30Hz Electroretinogram ( ERG) amplitude | Annual percent change per year at each of four years of followup
  Value in microvolts of response to 30hz ERG. Higher values = greater visual function
Change in Early Treatment of Diabetic Retinopathy(EDTRS) Visual Acuity | Change in number of letters read per year at each of four years of followup.
  Number of letters read per year. More letters read = better visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Eliot Berson (Deceased), MD, Principal Investigator — Berman-Gund Laboratory for the Study of Retinal Degenerations, Harvard Medical School
Locations (1):
- Berman-Gund Laboratory for the Study of Retinal Degenerations, Harvard Medical School, Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States

REFERENCES:
- [Background] Berson EL, Rosner B, Sandberg MA, Hayes KC, Nicholson BW, Weigel-DiFranco C, Willett W. A randomized trial of vitamin A and vitamin E supplementation for retinitis pigmentosa. Arch Ophthalmol. 1993 Jun;111(6):761-72. doi: 10.1001/archopht.1993.01090060049022. PMID 8512476
- [Result] Berson EL, Rosner B, Sandberg MA, Weigel-DiFranco C, Moser A, Brockhurst RJ, Hayes KC, Johnson CA, Anderson EJ, Gaudio AR, Willett WC, Schaefer EJ. Clinical trial of docosahexaenoic acid in patients with retinitis pigmentosa receiving vitamin A treatment. Arch Ophthalmol. 2004 Sep;122(9):1297-305. doi: 10.1001/archopht.122.9.1297. PMID 15364708
- [Result] Berson EL, Rosner B, Sandberg MA, Weigel-DiFranco C, Moser A, Brockhurst RJ, Hayes KC, Johnson CA, Anderson EJ, Gaudio AR, Willett WC, Schaefer EJ. Further evaluation of docosahexaenoic acid in patients with retinitis pigmentosa receiving vitamin A treatment: subgroup analyses. Arch Ophthalmol. 2004 Sep;122(9):1306-14. doi: 10.1001/archopht.122.9.1306. PMID 15364709
- [Derived] Comander J, Weigel DiFranco C, Sanderson K, Place E, Maher M, Zampaglione E, Zhao Y, Huckfeldt RM, Bujakowska KM, Pierce E. Natural history of retinitis pigmentosa based on genotype, vitamin A/E supplementation, and an electroretinogram biomarker. JCI Insight. 2023 Aug 8;8(15):e167546. doi: 10.1172/jci.insight.167546. PMID 37261916